CLINICAL TRIAL: NCT04195438
Title: Postoperative Heme Oxygenase Induction and Carbon Monoxide Production as a Novel Method to Assess Hepatic Regeneration and Predict Hepatic Related Morbidity After Partial Hepatectomy-1301GCC
Brief Title: Postoperative Heme Oxygenase Induction and Carbon Monoxide Production as a Novel Method to Assess Hepatic Regeneration and Predict Hepatic Related Morbidity After Partial Hepatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HP-00054854
Record Dates: First submitted 2019-11-20; First posted 2019-12-11 (Actual); Results first posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Liver Cancer
Keywords: Hepatectomy; Hepatic Regeneration; Arterial Blood Gas; CO Production
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Intervention Model Description: There is no randomization, every patient gets CO testing and ABG measurements to assess liver regeneration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Intervention Arm (Other): CO and ABG Testing Arm
  Interventions: Procedure: CO Testing Pre/Post Hepatic Resection; Diagnostic Test: ABG Testing Pre/Post Hepatic Resection; Diagnostic Test: CT Evaluations

INTERVENTIONS:
Procedure: CO Testing Pre/Post Hepatic Resection — Monitor CO in exhaled air of patients before liver resection, at 4 hours and 24 hours after PH
Diagnostic Test: ABG Testing Pre/Post Hepatic Resection — Monitor carboxyhemoglobin(COHb) in the arterial blood gas of patients before liver resection at 4 hours and 24 hours after PH
Diagnostic Test: CT Evaluations — Analyze the relationship between CO production and the extent of hepatic resection assessed by computed scans liver volumetric study at one and three months after PH, size and weight of the resected specimen and operative report

SUMMARY:
The study will monitor carbon monoxide production in patients undergoing liver resection. Carbon monoxide will be checked from arterial blood gas obtained routinely as a part of the postoperative care as well as from the exhaled air of the patient through a CO detector commercially available and used as smokerlyzer helping people to stop smoking. The results of the surgical resection will be collected from the patient routinely ordered tests after liver resection including pathology of the resected part of the liver, laboratory and radiology tests. The study aims to identify the relationship between CO production and recovery after liver resection. Results of this study may help in predicting and improving results of liver resection.

DETAILED DESCRIPTION:
The goal of this proposal is to elucidate the role of HO-1 induction in hepatic regeneration after partial hepatectomy (PH). There is a growing body of evidence that HO-1 induction through CO production has an important role in cellular protection and regeneration. To test this concept, we will monitor endogenous CO production in patients who undergo PH and analyze the relationship between CO production and hepatic regeneration. Using this approach we will test the following two hypotheses: (1) HO-1 induction after PH is proportional to the extent of the surgical resection, and (2) failure to appropriately induce HO-1 is associated with impaired hepatic regeneration.

Specific Aim 1: To monitor the extent of HO-1 induction (by measuring endogenous CO production) in relationship to the extent of hepatic resection 1.1 Monitor CO in exhaled air of patients before liver resection, at 4 hours and 24 hours after PH 1.2 Monitor carboxyhemoglobin(COHb) in the arterial blood gas of patients before liver resection at 4 hours and 24 hours after PH 1.3 Analyze the relationship between CO production and the extent of hepatic resection assessed by computed scans liver volumetric study at one and three months after PH, size and weight of the resected specimen and operative report.

Specific Aim 2: To analyze the relationship between HO-1 induction and the quality of post-hepatectomy liver regeneration after PH 2.1 Analyze the relationship between CO production and the quantity and quality of hepatic regeneration assessed by computed scans liver volumetric study at one and three months after PH and liver function tests after PH.

2.2 Determine the relation between postoperative liver related morbidity in patients undergoing PH and the extent of postoperative HO-1 induction.

ELIGIBILITY:
Inclusion Criteria:

* Patients plan to have partial liver resection for primary liver pathology or metastatic disease.
* Patients able to comprehend and willing to sign the written consent form.

Exclusion Criteria:

* Patients age less than 18
* Patients not having pathology proven liver malignancy
* Patient not able to comprehend or sign written consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-05-07 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cherif Boutros, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland Baltimore Washington Medical Center, Glen Burnie, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Aggregate data once data is analyzed and available when the study endpoints are completed patient enrollment is completed.
Supporting Information: Study Protocol, ICF
Time Frame: 12 months post study completion
Access Criteria: clinicaltrials.gov

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Arm
Started | 25
Completed | 24
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Intervention Arm
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 11
Age, Continuous [Median (Full Range); unit: years] | 64 [36 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: CO Output (Ppm)
Description: Measure HO-1 induction by measuring endogenous CO production in relationship to the extent of hepatic resection
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: ppm
Arm/Group | Intervention Arm
Number analyzed (Participants) | 24
ppm | 2.03 (0.82)

2. Primary Outcome: ABG (COHb)
Description: Measure HO-1 induction by measuring endogenous CO production in relationship to the extent of hepatic resection
Time Frame: Baseline
Measure: Mean (Full Range); unit: percentage of Carboxyhemoglobin
Arm/Group | Intervention Arm
Number analyzed (Participants) | 24
percentage of Carboxyhemoglobin | 1.58 [0.5 to 6.2]

3. Primary Outcome: CO Output (Ppm)
Description: Measure HO-1 induction by measuring endogenous CO production in relationship to the extent of hepatic resection
Time Frame: 4 hours post resection
Measure: Mean (Standard Deviation); unit: ppm
Arm/Group | Intervention Arm
Number analyzed (Participants) | 24
ppm | 3.11 (1.42)

4. Primary Outcome: ABG (COHb)
Description: Measure HO-1 induction by measuring endogenous CO production in relationship to the extent of hepatic resection
Time Frame: 4 hours post resection
Measure: Mean (Full Range); unit: percentage of Carboxyhemoglobin
Arm/Group | Intervention Arm
Number analyzed (Participants) | 24
percentage of Carboxyhemoglobin | 1.41 [0.4 to 2.8]

5. Primary Outcome: CO Output (Ppm)
Description: Measure the extent of HO-1 induction by measuring endogenous CO production in relationship to the extent of hepatic resection
Time Frame: 24 hours post resection
Measure: Mean (Standard Deviation); unit: ppm
Arm/Group | Intervention Arm
Number analyzed (Participants) | 24
ppm | 3.00 (1.41)

6. Primary Outcome: ABG (COHb)
Description: as for outcome 5
Time Frame: 24 hours post resection
Measure: Mean (Full Range); unit: percentage of Carboxyhemoglobin
Arm/Group | Intervention Arm
Number analyzed (Participants) | 24
percentage of Carboxyhemoglobin | 1.54 [0.9 to 2.3]

7. Secondary Outcome: Volume (ml)
Description: Measure the relationship between HO-1 induction and the quality of post-hepatectomy liver regeneration
Time Frame: One month after PH and liver function tests
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Intervention Arm
Number analyzed (Participants) | 24
ml | 170 (146)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Intervention Arm
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

LIMITATIONS AND CAVEATS:
Lower enrollment than planned Further studies will be necessary to identify patient and liver factors that influence the induction of HO-1 as well as its potential beneficial effect on liver regeneration and patient outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-21): https://cdn.clinicaltrials.gov/large-docs/38/NCT04195438/Prot_SAP_000.pdf